CLINICAL TRIAL: NCT03421288
Title: A Randomized, Open-label Phase II/III Efficacy and Safety Study of Atezolizumab in Combination With FLOT Versus FLOT Alone in Patients With Gastric Cancer and Adenocarcinoma of the Oesophago-gastric Junction and High Immune Responsiveness (MO30039/MO43340) - The IKF-DANTE Trial
Brief Title: Study of Atezolizumab + FLOT vs. FLOT Alone in Patients With GC/GEJ and High Immune Responsiveness
Acronym: DANTE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DANTE/FLOT8; 2017-001979-23 (EudraCT Number); MO30039/MO43340 (Other: Roche); AIO-STO-0317 (Other: AIO number); IKF-s633 (Other: Institut für Klinische Krebsforschung IKF)
Record Dates: First submitted 2018-01-11; First posted 2018-02-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — atezolizumab; Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: FLOT with Atezolizumab (Experimental): Patients randomized to treatment Arm A will receive atezolizumab (840 mg IV over 1 hour) + FLOT in four 2-week treatment cycles prior to undergoing surgery. Following surgery, patients will receive another four 2-week cycles of atezolizumab + FLOT followed by 8 additional 3-week treatment cycles with atezolizumab alone (maintenance setting: 1,200 mg q3w). FLOT can be deescalated to FLO, FLT or FL in case of chemorelated toxicity at any time and at the discretion of investigator.
  Interventions: Drug: Atezolizumab; Drug: 5-Fluorouracil; Drug: Calciumfolinat; Drug: Oxaliplatin; Drug: Docetaxel
- Arm B: FLOT alone (Active Comparator): Patients randomized to Arm B will receive FLOT alone for four 2-week treatment cycles prior to surgery. Following surgery, patients will receive another four 2-week cycles of chemotherapy alone. FLOT can be deescalated to FLO, FLT or FL in case of chemo-related toxicity at any time and at the discretion of investigator. Docetaxel 50 mg/m², d1 Oxaliplatin 85 mg/m², d1 Calciumfolinat 200 mg/m², d1 5-Fluorouracil 2600 mg/m², d1
  Interventions: Drug: 5-Fluorouracil; Drug: Calciumfolinat; Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Atezolizumab — Day 1 q2w: 840 mg IV over 1 hour (4 cycles perioperative with FLOT) + Day 1 q3w: 1200 mg IV over 1 hour (8 additional cycles monotherapy)
  Other Names: TECENTRIQ
  Arms: Arm A: FLOT with Atezolizumab
Drug: 5-Fluorouracil — Day 1 q2w: 2600 mg/m² IV over 24 hours
  Other Names: 5-FU
Drug: Calciumfolinat — Day 1 q2w: 200 mg/m² IV over 1 hour
  Other Names: Leucovorin
Drug: Oxaliplatin — Day 1 q2w: 85 mg/m² IV over 2 hours
  Other Names: ELOXATIN
Drug: Docetaxel — Day 1 q2w: 50 mg/m² IV over 1 hour
  Other Names: TAXOTERE

SUMMARY:
This is a multicenter, randomized, controlled, open-label study comparing perioperative atezolizumab with FLOT chemotherapy versus FLOT alone in patients with locally advanced, operable adenocarcinoma of the stomach or GEJ with high immune responsiveness.

DETAILED DESCRIPTION:
The study will evaluate the safety and efficacy of the study treatment regimens. Potential study participants will be assessed for eligibility during a 28-day screening period. Only immune-competent patients with either of the following MSI-high, PD-L1 CPS≥1, TMB ≥10/MB or EBV+ will be enrolled. Eligible patients will be randomized to perioperative treatment with either atezolizumab with FLOT (Arm A) or FLOT alone (Arm B). Randomization will occur in a 1:1 ratio with stratification by clinical nodal stage (N+ vs. N-), location of the primary (GEJ type I vs. GEJ type II/III vs. stomach), and PD-L1-combined positive score (CPS≥5 vs. CPS<5) or MSI-status (MSI/MMRd vs. MSS/MMRp).

Following randomization, study patients will enter the study treatment period which will last approximately 22 to 52 weeks depending on treatment arm and timing of surgery.

Arm A: FLOT with Atezolizumab:

Patients randomized to treatment Arm A will receive atezolizumab + FLOT in four 2-week treatment cycles as described below prior to undergoing surgery. Following surgery, patients will receive another four 2-week cycles of atezolizumab + FLOT followed by 8 additional 3-week treatment cycles with atezolizumab alone.

Arm B: FLOT alone:

Patients randomized to Arm B will receive FLOT alone for four 2-week treatment cycles prior to surgery. Following surgery, patients will receive another four 2-week cycles of chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. In the investigator's judgement, is willing and able to comply with the study protocol including the planned surgical treatment
3. Female and male patients* ≥ 18 years of age
4. Diagnosed with histologically confirmed adenocarcinoma of the GEJ (Type I-III) or the stomach (cT2, cT3, cT4, any N category, M0), or (any T, N+, M0) that:

   1. is not infiltrating any adjacent organs or structures by CT or MRI evaluation
   2. does not involve peritoneal carcinomatosis
   3. is considered medically and technically resectable Note: the absence of distant metastases must be confirmed by CT or MRI of the thorax and abdomen, and, if there is clinical suspicion of osseous lesions, a bone scan. If peritoneal carcinomatosis is suspected clinically, its absence must be confirmed by laparoscopy. Diagnostic laparoscopy is mandatory in patients with T3 or T4 tumors of the diffuse type histology in the stomach.
5. No prior cytotoxic or targeted therapy
6. No prior partial or complete esophagogastric tumor resection
7. ECOG ≤ 1
8. Phase II only: Availability of a representative tumor specimen that is suitable for determination of PD-L1 and MSI status; MSI assessment will be performed locally or centrally, and result must be available prior to randomization (for details, see chapter 9.1). PD-L1 will be assessed centrally but is not used for enrolment of the patients. The analysis requires paraffin embedded biopsy samples of the tumor.

   Phase III only: Assessment of MSI and PD-L1 [and optional TMB/EBV] must be performed locally and results for either of the following MSI-high, PD-L1 CPS≥1, TMB ≥10/MB or EBV+ must be available prior to randomization (for details, see chapter 9.2).
9. Females of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 5 months after the last study treatment. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (has not had ≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal implants, established, proper use of combined oral or injected hormonal contraceptives, and certain intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

   Males must agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agree to refrain from donating sperm, as defined below:

   a. With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of 1% per year during the treatment period and for at least 3 months after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period. Men with a pregnant partner must agree to remain abstinent or to use a condom for the duration of the pregnancy.
10. Criterion integrated in criterion 9.
11. Adequate hematological, hepatic and renal function as indicated by the following parameters:

    * Leukocytes ≥ 3.000/mm³, platelets ≥ 100.000/mm3without transfusion, absolute neutrophil count (ANC) ≥ 1500/mm3without granulocyte colony-stimulating factor support, Hemoglobin ≥ 90 g/L (9 g/dL) - Patients may be transfused to meet this criterion.
    * Bilirubin ≤ 1.5 x upper limit of normal, aspartate transaminase and alanine transaminase ≤ 2.5 x upper limit of normal, alkaline phosphatase ≤ 2.5 x upper limit of normal
    * Serum creatinine ≤ 1.5 x upper limit of normal, or glomerular filtration rate > 45 ml/min (calculated using the Cockcroft-Gault formula)
    * Serum albumin ≥ 25 g/L (2.5 g/dL)
    * For patients not receiving therapeutic anticoagulation: INR or aPTT ≤ 1.5 x ULN; for patients receiving therapeutic anticoagulation: stable anticoagulant regimen *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.

Exclusion Criteria:

1. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein; Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
2. Any known contraindication (including hypersensitivity) to docetaxel, 5-FU, leucovorin, or oxaliplatin.
3. Active or History of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone, or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible based on consultation with the sponsor's medical monitor. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

   * Rash must cover < 10% of body surface area
   * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
   * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
4. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
5. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, idiopathic pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan.

   Note: History of radiation pneumonitis within the radiation field (fibrosis) is permitted.
6. Positive test for human immunodeficiency virus (HIV)
7. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen antibody test) are eligible. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction testing is negative for HCV ribonucleic acid (RNA).
8. Active tuberculosis
9. Known dihydropyrimidine dehydrogenase (DPD) deficiency. Patients with a reduced DPD activity (CPIC activity score of 1.0-1.5) might participate in the study and receive a reduced dosage of 5-FU after discussion with the lead investigator and sponsor
10. Uncontrolled tumor-related pain; Patients requiring pain medication must be on a stable regimen at study entry
11. Administration of a live, attenuated vaccine within four weeks prior to start of enrollment, or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after the last dose of atezolizumab
12. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibodies
13. Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within four weeks or five half-lives of the drug, whichever is longer, prior to study enrollment
14. Treatment with systemic corticosteroids or other systemic immunosuppressive medications within 2 weeks prior to study enrollment. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
15. Significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to initiation of study treatment, unstable arrhythmias, or unstable angina.
16. Clinically significant valvular defect
17. History of other malignancy within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g. 5-year OS rate >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ or Stage I uterine cancer
18. Known central nervous system metastases
19. Peripheral polyneuropathy ≥ NCI CTCAE grade 2
20. Serum albumin < 2.5 g/dL.
21. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
22. Serious infection requiring oral or IV antibiotics within 14 days prior to study enrollment
23. Chronic inflammatory bowel disease
24. Clinically significant active gastrointestinal bleeding
25. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment
26. Evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results
27. Participation in another interventional clinical study ≤ 30 days prior to study enrollment or planned participation in such a study at the same time as this study
28. Receipt of an investigational drug within 28 days prior to initiation of study drug
29. Pregnancy or breast feeding or planning to become pregnant within 5 months after the end of treatment. Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Event free survival (EFS) between arms | 10 years
  to compare Event free survival (EFS) in patients with locally advanced, operable esophagogastric adenocarcinoma receiving perioperative FLOT with atezolizumab versus FLOT alone in the intent to treat population (ITT) and where EFS is defined as the time from randomization to disease progression or relapse after surgery or death from any cause

SECONDARY OUTCOMES:
Pathological complete regression (pCR, TRG 1a by Becker) rate | after 4 cycles (each cycle is 14 days) + surgery; i.e. after 12 weeks in total
  Pathological complete regression (pCR, TRG 1a by Becker) rate where pCR is defined as the absence of residual tumor based on evaluation of the resected esophagogastric specimen in the primary by a central reference pathologist
Pathological complete and subtotal regression (TRG1a/b by Becker) | after 4 cycles (each cycle is 14 days) + surgery; i.e. after 12 weeks in total
  Pathological complete and subtotal regression (TRG1a/b by Becker). TRG1a/b is defined as < 10% residual tumor per tumor bed based on evaluation of the resected esophagogastric specimen in the primary by a central reference pathologist.
R0 resection rate | after 4 cycles (each cycle is 14 days) + surgery; i.e. after 12 weeks in total
  R0 resection rate where R0 resection is defined as a microscopically margin negative resection with no gross or microscopic tumor remains in the areas of the primary tumor and/or sampled regional lymph nodes based on evaluation by the local pathologist.
Overall survival (OS) | 10 years
  Overall survival (OS) where OS is defined as the time from randomization to death from any cause
Overall survival (OS) and EFS in the subgroup of patients with PD-L1 CPS score ≥ 5 and ≥ 10 and patients with MSI | 10 years
  Overall survival (OS) where OS is defined as the time from randomization to death from any cause and EFS, where EFS is defined as the time from randomization to disease progression or relapse after surgery or death from any cause, both compared between the specific subgroups

OTHER OUTCOMES:
Detectable ctDNA after curative surgery | after surgery (approx. 12 weeks after first dose)
  Prevalence of detectable ctDNA in patients after curative surgery
ctDNA clearance on treatment | at baseline, before and after surgery (approx. 10 and 12 weeks after first dose), during study treatment (for up to 1 year), in case of relaps/progression
  Cumulative incidence of ctDNA clearance (on treatment) compared between arms

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Study Director — Institute of Clinical Cancer Research IKF at Krankenhaus Nordwest; Thorsten Goetze, Prof., Principal Investigator — University Cancer Center Frankfurt, Krankenhaus Nordwest
Locations (2):
- Krankenhaus Nordwest, Frankfurt, Germany
- SAKK Coordinating Center, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Lorenzen S, Gotze TO, Thuss-Patience P, Biebl M, Homann N, Schenk M, Lindig U, Heuer V, Kretzschmar A, Goekkurt E, Haag GM, Riera-Knorrenschild J, Bolling C, Hofheinz RD, Zhan T, Angermeier S, Ettrich TJ, Siebenhuener AR, Elshafei M, Bechstein WO, Gaiser T, Loose M, Sookthai D, Kopp C, Pauligk C, Al-Batran SE; AIO and SAKK Study Working Groups. Perioperative Atezolizumab Plus Fluorouracil, Leucovorin, Oxaliplatin, and Docetaxel for Resectable Esophagogastric Cancer: Interim Results From the Randomized, Multicenter, Phase II/III DANTE/IKF-s633 Trial. J Clin Oncol. 2024 Feb 1;42(4):410-420. doi: 10.1200/JCO.23.00975. Epub 2023 Nov 14. PMID 37963317
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069